CLINICAL TRIAL: NCT02018432
Title: Adherence to Therapy in COPD Patients Under Dose Escalation of Roflumilast
Brief Title: Strategy to Improve Adherence of Roflumilast
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sei Won Lee, Department of Pulmonary and Critical Care Medicine and Clinical Research Center for Chronic Obstructive Airway Diseases, Asan Medical Center, University of Ulsan College of Medicine, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Roflumilast_compliance
Record Dates: First submitted 2013-12-12; First posted 2013-12-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Roflumilast escalation dosage (Experimental): Roflumilast 250 μg qd (4 weeks) →500 μg qd
  Interventions: Drug: Roflumilast escalation dosage
- Roflumilast conventional dosage (Experimental): Roflumilast 500 μg qd
  Interventions: Drug: Roflumilast conventional dosage

INTERVENTIONS:
Drug: Roflumilast escalation dosage — This is a randomized, prospective, open label, comparative study to assess whether the administration of roflumilast by dose escalation varies the incidence of discontinuations due to adverse events when compared with the usual dosage in severe and very severe COPD patients.
  Roflumilast 250 μg once daily for 4 weeks and then increased dose of Roflumilast 500 μg once daily for 12 weeks
  Other Names: Daxas
  Arms: Roflumilast escalation dosage
Drug: Roflumilast conventional dosage — Roflumilast 500 μg once daily for 12 weeks
  Other Names: Daxas
  Arms: Roflumilast conventional dosage

SUMMARY:
Main adverse events of Roflumilast are weight loss, loss of appetite, insomnia, headache, diarrhea, vomiting, and nausea. Although the majority of these adverse reactions were mild or moderate. They occurred mainly at the beginning of therapy and mostly resolved with continued treatment around for two weeks according to experiences of clinicians. These adverse events occur more often in Roflumilast 500 μg than 250 μg, having negative impact on compliance of patients at the early stage of treatments.

Thus, investigators aim to compare the drop-out rates between the usual dosage (Roflumilast 500 μg once daily) and the dose escalation (Roflumilast 250 μg once daily for 4 weeks and then escalating dose of 500 μg once daily).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female older than 40 years
2. Clinical diagnosis of COPD (confirmed with a post-bronchodilator forced expiratory volume in 1 s [FEV1]/forced vital capacity [FVC] ratio ≤70%) at least 4 weeks prior to the study and post-bronchodilator FEV1 is 50% or less than the predicted value
3. Former smokers or current smokers with at least a 10 pack-year history
4. A history of exacerbation (scheduled/unscheduled visits to primary care physicians, specialists or allied healthcare professionals, or emergency room, or hospitalization due to purulent sputum or increased sputum, or increased dyspnea) in the previous year (at least one)
5. Chronic bronchitis (cough and sputum production for at least three months within two years)
6. Able to have the signed written informed consent prior to any study-related procedures.

Exclusion Criteria:

1. COPD exacerbation or respiratory infection 4 weeks prior to the baseline visit
2. Known a1-antitrypsin deficiency
3. Need for long-term oxygen therapy
4. Moderate to severe liver impairment (Child-Pugh B or C)
5. Severe immunological diseases (e.g. HIV infection, multiple sclerosis, lupus erythematosus, etc)
6. Severe acute infectious diseases
7. Cancers
8. Subjects being treated with immunosuppressive medicinal products (i.e.: methotrexate, azathioprine, infliximab, etanercept, or oral corticosteroids to be taken long-term) except short-term systemic corticosteroids)
9. Latent infections such as tuberculosis, viral hepatitis, herpes viral infection and herpes zoster
10. Subjects with congestive heart failure (NYHA grades 3 and 4)
11. Subjects with a history of depression associated with suicidal ideation or behavior
12. Clinically meaningful bronchiectasis
13. Pregnancy or breast feeding, or Female subjects of childbearing potential unwilling to use effective contraception
14. Patients with known hypersensitivity to Roflumilast or rescue medication and their ingredients
15. Patients with previous Roflumilast therapy within past 3 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
medication(Roflumilas) history taking | 16 weeks
  In every follow-up, patients will be asked about their medication history. The patients will count the rest of the Roflumilast that they are going to take in the future.

SECONDARY OUTCOMES:
Laboratory test : Hematology, Biochemistry, and Urinalysis | 16 weeks
  •Laboratory test : Hematology, Biochemistry, and Urinalysis
Urine pregnancy test | 16 weeks
  •Urine pregnancy test
Chest X-ray Test | 16 weeks
  •Chest X-ray Test
ECG Test | 16 weeks
  •ECG Test
Lung Function Test | 16 weeks
  •Lung Function Test
QoL Questionnaire (CAT score) | 16 weeks
  •QoL Questionnaire (CAT score)
Other tests (HBsAg, HCV, HIV) | 16 weeks
  •Other tests (HBsAg, HCV, HIV)

CONTACTS AND LOCATIONS:
Overall Officials: Sei Won Lee, MD, Principal Investigator — Department of Pulmonary and Critical Care Medicine and Clinical Research Center for Chronic Obstructive Airway Diseases, Asan Medical Center, University of Ulsan College of Medicine, Seoul, Republic of Korea
Locations (1):
- Department of Pulmonary and Critical Care Medicine and Clinical Research Center for Chronic Obstructive Airway Diseases, Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Park TS, Kang J, Lee JS, Oh YM, Lee SD, Lee SW. Adherence to roflumilast under dose-escalation strategy in Korean patients with COPD. Int J Chron Obstruct Pulmon Dis. 2019 Apr 16;14:871-879. doi: 10.2147/COPD.S191033. eCollection 2019. PMID 31354255